CLINICAL TRIAL: NCT04178018
Title: Transvaginal Ultrasound and Photoacoustic Imaging of the Ovary
Brief Title: Transvaginal Ultrasound and Photoacoustic Imaging of Ovary
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201608016-2; 1R01CA237664-01A1 (NIH)
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Ovary; Anomaly
MeSH Terms: conditions — Congenital Abnormalities | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Transvaginal photoacoustic imaging/ultrasound (Experimental): * Baseline transvaginal ultrasound (standard of care) followed by transvaginal ultrasound and photoacoustic imaging for all participants enrolled
  * Once the surgeon has surgically removed the ovary(ies), they will be imaged with the photoacoustic imaging/ultrasound
  * For the exploratory outcome measure for high risk participants (approximately 50 participants), the transvaginal ultrasound (standard of care) followed by transvaginal ultrasound and photoacoustic imaging will be performed additionally at 6 months, 12 months, 18 months, 24 months, and at the time of surgery
  * For the exploratory outcome measure for high risk participants (approximately 10 participants), the transvaginal ultrasound (standard of care) followed by transvaginal ultrasound and photoacoustic imaging will be performed additionally every 2 weeks at follicular phase and at the luteal phase for 3 months
  Interventions: Device: Photoacoustic imaging; Device: Ultrasound

INTERVENTIONS:
Device: Photoacoustic imaging — -Emerging technique in which a short-pulsed laser beam penetrates diffusively into a tissue sample
  Other Names: PAI; Photoacoustic tomography
Device: Ultrasound — -The ultrasound is being used in conjunction with the photoacoustic imaging

SUMMARY:
This study is being conducted to validate if photoacoustic imaging potentially reduces benign surgeries without compromising cancer detection sensitivity. The study will also explore whether using the photoacoustic imaging/ultrasound technique has any potential with early ovarian cancer detection in a group of high risk patients.

DETAILED DESCRIPTION:
In primary and secondary objectives, the investigators will consent patients who are at risk for ovarian cancer, or who have an ovarian mass possibly suggestive of a malignancy and are counseled to undergo oophorectomy. Patients will be identified by the GYN physicians and consented by the study coordinator prior to the date of the scheduled surgical procedure.

In exploratory objectives, the investigators will consent patients who are at risk for ovarian cancer and wish to be followed before making decision to undergo prophylactic oophorectomy. Patients will be identified based on the eligibility criteria by the physicians and consented by the study coordinator prior to the follow up studies.

ELIGIBILITY:
Inclusion Criteria for Primary and Secondary Outcome Measures

* All patients, 18 years or older, referred to the Washington University School of Medicine for conditions necessitating surgery to include at least a unilateral oophorectomy.
* Willingness to participate in the study and able to provide informed consent.

Inclusion Criteria for Exploratory Outcome Measures

* At least 18 years of age
* Referred to the Washington University School of Medicine for conditions necessitating surgery to include at least a unilateral oophorectomy, an ovarian cystectomy, or a unilateral or bilateral salpingectomy .
* Willing to be followed for one to 4.5 years prior to making the decision to undergo prophylactic oophorectomy.
* Documented deleterious mutation in one of the following ovarian cancer genes: BRCA1, BRCA2, BRIP1, PALB2, RAD51C, RAD51D, BARD1, MSH2, MSH6, MLH1, PMS2, or EPCAM.

Exclusion Criteria:

* Male
* Younger than 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2020-02-09 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Assess the impact of co-registered PAI/US on the potential reduction of benign surgeries as measured by the area under receiver characteristic curve (AUC) | At the time of surgery (estimated to be 2 weeks)
  The anticipated improvement of diagnostic accuracy on reduction of surgeries of benign ovaries will be from current practice of AUC=55% to AUC=78%.

SECONDARY OUTCOMES:
False negative rate of conventional imaging compared to conventional imaging & PAI/US as measured by sensitivity of cancer detection | At the time of surgery (estimated to be 2 weeks)
  The anticipated improvement of cancer detection accuracy will be from current practice of 80% to 94%.

OTHER OUTCOMES:
Determine if co-registered PAI/US can be used as a sensitive and specific screening tool for early detection of malignant neoangiogenesis within a group of high-risk women | Through completion of follow-up (estimated to be 4.5 years)
  The investigators hope to improve current practice by detecting early cancers from this group of high-risk women
Determine normal changes of photoacoustic imaging parameters | Through completion of follow-up (estimated to be 4.5 years)
  The investigators expect to see small changes of the PAI/US imaging parameters of less than 10-15 for repeated measurements of 3 menstrual cycles

CONTACTS AND LOCATIONS:
Overall Officials: Cary L Siegel, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing of data collected by this project is essential to gain knowledge on how to improve and manage the current standard of care on high-risk and ovarian cancer patients.
  The investigators will share data through multiple channels including:
  * Publication of results and findings at various stages in peer-reviewed journals
  * Presentation of results and findings at national and international conferences
  * Public access to data collected from this project upon reasonable request when the study is completed.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu